CLINICAL TRIAL: NCT03850899
Title: Alcoholic Hepatitis Network Observational Study
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Samer Gawrieh, Co-Director, Alcoholic Hepatitis Network Data Coordinating Center and Associate Professor of Medicine Division of Gastroenterology and Hepatology, Indiana University
Other Study IDs: AlcHepNet-01
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: Heavy drinkers with alcoholic hepatitis
- Controls: Heavy drinkers without significant liver disease
- Donor: Healthy non-drinkers

SUMMARY:
The purpose of this research study is to create a clinical database and bio-repository. To do this, we will obtain blood, urine, saliva, and stool samples (e.g., biological samples) and personal health information from you to use in future research studies related to alcoholic hepatitis or other diseases. Part of your blood sample will be used to extract your DNA. DNA is the genetic material that gives us unique characteristics. We are doing this research study because we are trying to find out more about how and why illnesses related to alcoholic hepatitis or other diseases occur in people. To do this, we will study the biological samples and personal health information from healthy and sick people.

A "biological sample" is usually blood, but can be any body fluid. "Personal Health Information" includes such items as your name, age, gender, race, and/or your medical information. It can also include data from measurements and tests that you had while participating in another research study or that were done during the course of your regular medical care or doctor visits.

DETAILED DESCRIPTION:
What should I know about this research?

* Someone will explain this research to you.
* Taking part in this research is voluntary. Whether you take part is up to you.
* If you don't take part, it won't be held against you.
* You can take part now and later drop out, and it won't be held against you
* If you don't understand, ask questions.
* Ask all the questions you want before you decide.

How long will I be in this research? We expect that your taking part in this research will last up to 6 months, after the 6 months we will look in your medical records every 180 days for up to five years.

Why is this research being done? The purpose of this research is to create a clinical database and bio-repository to study alcoholic hepatitis.

What happens to me if I agree to take part in this research? If you decide to take part in this research study, the general procedures include: 1) allowing the investigators to review your medical records, 2) answering questions about you and your health, 3) completing questionnaires about alcohol use, 4) having a physical exam and blood drawn, and 5) providing urine and stool samples.

Could being in this research hurt me? The most important risks or discomforts that you may expect from taking part in this research include mild pain from blood draws and a small chance for a loss of confidentiality (e.g., unauthorized users gain access to sensitive and protected data about you).

Will being in this research benefit me? It is not expected that you will personally benefit from this research. Possible benefits to others may include understanding specific health conditions in patients with alcoholic hepatitis or other diseases.

ELIGIBILITY:
CASES: Heavy drinkers with alcoholic hepatitis

Inclusion criteria

1. A clinical diagnosis of alcoholic hepatitis as defined by the NIAAA pan-consortia for AH:

   1. Onset of jaundice (defined as serum total bilirubin >3 mg/dL) within the prior 8 weeks to screening visit
   2. Regular consumption of alcohol with an intake of > 40 gm daily or >280gm weekly on average for women and > 60 gm daily or >420gm weekly on average for men for 6 months or more, with less than 8 weeks of abstinence before onset of jaundice
   3. AST > 50 IU/l
   4. AST:ALT > 1.5 and both values < 400 IU/l
   5. and/or histological evidence of AH*
2. Serum total bilirubin >3 mg/dL
3. Subject or guardian ability to understand and willingness to provide written consent
4. Age greater or equal to 21 years
5. Re-enrolment of an alcoholic hepatitis donor is permissible up to 4 times if the donor presents with a new episode of alcoholic hepatitis 24 weeks or longer after the most recent enrolment in the study

Exclusion criteria

1. Liver disease significantly caused by hemochromatosis, autoimmune liver disease, Wilson disease, and acute viral hepatitis (NOTE: The presence of chronic hepatitis C, hepatitis B, HIV, or stage 1 (one lesion <2 cm) HCC is not exclusion to participation)
2. Pregnant or breast feeding
3. Received liver transplant
4. Based on the judgment of the investigator, subject is not capable of understanding or complying with the study requirements

CONTROLS: Heavy drinkers without significant liver disease Inclusion criteria

1. History of chronic alcohol consumption sufficient to cause liver damage. Generally, this is considered to be >40 g/day or >280g/week on average for women and >60 g/day or >420 g/week on average for men, for 6 months or more. Judgement about chronic alcohol consumption will be made by the site investigator.
2. Subject or guardian ability to understand and willingness to provide written consent
3. Age greater or equal to 21 years

Exclusion criteria

1. Past evidence of alcoholic liver disease, defined as a bilirubin > 2.0 mg/dL, an AST > 1.5 ULN, and any hospital admission for liver disease, or the presence of esophageal varices or ascites (at any time in the past)
2. Liver disease significantly caused by hemochromatosis, autoimmune liver disease, Wilson disease, NAFLD, and acute viral hepatitis (NOTE: The presence of chronic hepatitis C, hepatitis B, or HIV is not exclusion to participation.)

   *Individuals with a diagnosis of Gilbert's can have total bilirubin up to 3.0 mg/dL and still be eligible for participation.
3. Alcohol intake at less than 40 g/day or 280g/week on average for women and 60 g/day or 420 g/week on average for men for longer than the past 28 days
4. If liver stiffness has been assessed within the prior 90 days, then stiffness suggesting fibrosis of F1 or greater is excluded. For Fibroscan, this is a fibrosis score >7.0 kPa.
5. Received liver transplant
6. Pregnant or breast feeding
7. Any of the following laboratory abnormalities within 90 days prior to signing the consent.

   1. Total bilirubin: >ULN*
   2. INR: > 1.4

Healthy Controls

Inclusion criteria

1. AUDIT-C scores of <4 for men and <3 for women (signifying no alcohol misuse)
2. Abstinent (consumption of less than one standard drink/week) during the 6 months prior to enrolment
3. Ability to understand and willingness to provide written consent.
4. Age greater or equal to 21 years

Exclusion criteria

1. Clinical history or laboratory evidence of liver disease including alcoholic liver disease, NAFLD, hemochromatosis, alcoholic hepatitis, autoimmune liver disease, Wilson disease, hepatitis C, or hepatitis B.
2. Presence of diabetes (requiring treatment with oral agents or insulin).
3. Significant heart disease (prior history of heart disease, other than hypertension)
4. Chronic lung disease (requiring chronic treatment)
5. Immune related conditions (such as Crohn's disease, rheumatoid arthritis, ulcerative colitis, systemic lupus erythematosus, severe psoriasis, etc.)
6. Known infection with HIV
7. Presumed infection, or use of antibiotics or other medications (e.g., corticosteroids) that would affect immune function, within the past 14 days
8. BMI>35
9. Current or known history of cancer (except in situ carcinoma of the cervix or adequately treated basal or squamous cell carcinoma of the skin) within 5 years prior to enrollment
10. Received liver transplant
11. Pregnant or breast feeding
12. Any of the following laboratory abnormalities within 90 days prior to signing the consent.

    1. Hemoglobin: <10 g/dL
    2. Conjugated bilirubin: > ULN
    3. INR: > 1.4
    4. AST: >40 IU/mL
    5. ALT: >40 IU/mL
13. Based on the judgment of the investigator, subject is not capable of complying with the study requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any subject with Alcoholic hepatitis, Heavy healthy drinkers, and Healthy controls
Sampling Method: Probability Sample
Enrollment: 1133 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - IU School of Medicine, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University Of Massachusetts, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical School, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dasarathy S, Tu W, Bellar A, Welch N, Kettler C, Tang Q, Liangpunsakul S, Gawrieh S, Radaeva S, Mitchell M; AlcHepNet. Development and evaluation of objective trial performance metrics for multisite clinical studies: Experience from the AlcHep Network. Contemp Clin Trials. 2024 Mar;138:107437. doi: 10.1016/j.cct.2024.107437. Epub 2024 Jan 11. PMID 38215876

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cases | Controls | Donor
Started | 717 | 257 | 159
Completed | 230 | 118 | 159
Not Completed | 487 | 139 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Donor | Total
Number analyzed (Participants) | 717 | 257 | 159 | 1133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 694 | 229 | 156 | 1079
  >=65 years | 23 | 28 | 3 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 294 | 109 | 99 | 502
  Male | 423 | 148 | 60 | 631
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 7 | 16 | 86
  Not Hispanic or Latino | 638 | 247 | 140 | 1025
  Unknown or Not Reported | 16 | 3 | 3 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 0 | 10
  Asian | 4 | 0 | 27 | 31
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 82 | 64 | 18 | 164
  White | 601 | 183 | 101 | 885
  More than one race | 4 | 2 | 3 | 9
  Unknown or Not Reported | 20 | 2 | 9 | 31
Region of Enrollment [Number; unit: participants]
  United States | 717 | 257 | 159 | 1133

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Clinical Data Collected
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls | Donor
Number analyzed (Participants) | 717 | 257 | 159
Participants | 717 | 257 | 159

2. Secondary Outcome: Number of Subjects With Bio-samples Collected
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls | Donor
Number analyzed (Participants) | 717 | 257 | 159
Participants | 698 | 247 | 159

ADVERSE EVENTS:
Time Frame: 5 years, 2 months
Arm/Group | Cases | Controls | Donor
All-Cause Mortality (participants affected / at risk) | 194/717 | 4/257 | 0/159
Serious Adverse Events (participants affected / at risk) | 0/717 | 0/257 | 0/159
Other Adverse Events (participants affected / at risk) | 0/717 | 0/257 | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03850899/Prot_SAP_000.pdf